CLINICAL TRIAL: NCT06556160
Title: Basic and Clinical Studies of Cochlear Synaptopathy
Brief Title: Fundamental and Clinical Study of Cochlear Synaptopathy
Acronym: FunCoSy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PO23045
Record Dates: First submitted 2023-08-17; First posted 2024-08-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hearing Loss
Keywords: Hearing Loss; Deafness; Micro vascular decompression; otoneurosurgery; retrosigmoid approach
MeSH Terms: conditions — Hearing Loss; Deafness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hearing impaired patients (Experimental): have a sensorineural hearing loss defined by hearing thresholds of 20 dB HL or better from 0.25 to 2 kHz and from 20 dB HL excluded to 55 dB HL at frequencies above 2 kHz.
  Interventions: Procedure: near field recording of human auditory nerve activity during retro sigmoid approach with contact electrode
- normal hearing patients (Active Comparator): free of neuro-sensory deafness, defined by mean hearing thresholds of less than or equal to 20 dB HL in pure tone audiometry in air conduction bilaterally on the side of the ear operated on and on the non-operated side from 0.25 to 8 kHz
  Interventions: Procedure: near field recording of human auditory nerve activity during retro sigmoid approach with contact electrode

INTERVENTIONS:
Procedure: near field recording of human auditory nerve activity during retro sigmoid approach with contact electrode — During surgery using a retro-sigmoid approach in the cerebellopontine angle (microvascular decompression), near-field recording of human auditory nerve activity using a contact electrode is performed on patients with normal or impaired hearing threshold.
  Each patient is explored preoperatively by hearing tests to search synaptopathie. During the surgery, stimuli are delivered.

SUMMARY:
In humans, surface electrophysiological recording of the cochlear nerve in response to a sound stimulus provides information about the integrity and function of synapses (synaptic transmission) and nerve fibre function. However, this information remains global. The investigators have preliminary data showing that it is possible to extract and characterise the functional properties of nerve fibres during otoneurosurgery in humans, and therefore to isolate the neuronal sub-populations mentioned above more precisely than is currently possible. The use of these electrophysiological data from near-field recordings, i.e. in contact with the nerve, will enable the design and improvement of a mathematical model of the human cochlea. This model will provide access to the individual responses of each nerve fibre and fill the current gap in knowledge between the functioning of these fibres and global surface recordings.

DETAILED DESCRIPTION:
During functional surgery on the cerebellopontine angle, a ball electrode is placed on the human cochlear nerve to monitor hearing. Once the electrode is in place, clicks and random noise bands will be delivered in order to analyze the cochlear electrophysiological signal produced. Depending on the characteristics recorded, this signal can be used at a given frequency and intensity to identify the populations of auditory neurons mainly involved. Prior to surgery, each patient will have been examined by the audiologist in order to determine the auditory thresholds in silence and noise, in tone and in speech, to carry out the digit test and to perform an electrocochleography and distortion products. Each result analyzed will be the subject of a further analysis using the mathematic model of the human cochlea.

ELIGIBILITY:
inclusion criteria :

Patients with normal hearing will be included:

* male or female
* over 18 and up to 70 years of age
* normal otoscopic examination
* due to undergo surgery on the cerebellopontine angle (microvascular decompression).
* free of neuro-sensory deafness, defined by mean hearing thresholds of less than or equal to 20 dB HL in pure tone audiometry in air conduction bilaterally on the side of the ear operated on and on the non-operated side from 0.25 to 8 kHz
* affiliated to a social security scheme
* have read the information note describing the study and have agreed in writing to take part by signing the informed consent form.

Patients with a hearing impairment will be included:

* male or female
* over 18 and up to 70 years of age
* normal otoscopic examination
* due to undergo surgery on the cerebellopontine angle (microvascular decompression).
* have a sensorineural hearing loss defined by hearing thresholds of 20 dB HL or better from 0.25 to 2 kHz and from 20 dB HL excluded to 55 dB HL at frequencies above 2 kHz.
* have read the information note describing the study and have agreed in writing to take part by signing the informed consent form.

exclusion criteria :

- Patients will be excluded from the study for whom the auditory nerve is not accessible during surgery, in particular because of complete tumour invasion of the cochlear nerve (stage III and IV neuroma, advanced meningioma) or because of a particular anatomical feature not identified during the preoperative examination, making it impossible to expose the nerve for recordings (protrusion of the posterior surface of the rock).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
In response to a stimulus, the neurophonic potential recorded in the form of a wave called PSTR will be characterised patients defined as normo and hearing loss based on preoperative audiometric tests | At 48 months
  During ponto cerebellum retro sigmoide surgery. In response to a stimulus, the neurophonic potential recorded in the form of a wave called PSTR will be characterised patients defined as normo and hearing loss based on preoperative audiometric tests by the following indices:- the amplitude of the peak- the amplitude of the plateau- the peak to plateau ratio- the time constant for the rapid decay of the peak- the time constant for the slow decay of the peak.
Compare the amplitude and spectrum of global evoked auditory nerve activity with basic stimuli between patients defined as normo and hearing loss based on preoperative audiometric tests | At 48 months
  During ponto cerebellum retro sigmoide surgeryelectrocochleography and distortion products.

SECONDARY OUTCOMES:
compare the primary objective with the results obtained with a mathematical model of the human cochlea in order to improve the responses of our model. | At 48 months
  During ponto cerebellum retro sigmoide surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France